CLINICAL TRIAL: NCT00916084
Title: This Study is to Apply the Tongue Force to Correct the Dentofacial Deformities
Brief Title: Comparative Results of Maxillary Deficiency Treatment by Fixed Tongue Appliance and Fixed Facemask in Growing Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University (Other)
Responsible Party: Shahid Beheshti Medical University, Shahid Beheshti Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: behnaz1357
Record Dates: First submitted 2009-06-08; First posted 2009-06-09 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2009-12

CONDITIONS: Maxillary Deficiency
MeSH Terms: conditions — Retrognathia | interventions — Masks

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental)
  Interventions: Device: Fixed Tongue Appliance
- Group B (Experimental)
  Interventions: Device: Fixed Face Mask

INTERVENTIONS:
Device: Fixed Tongue Appliance — A functional appliance used for maxillary protraction. It has two bands on first molars, expansion screw and long palatal plate in the canine area which cages the tongue and transfers the force of the tongue during physiological activity to the upper arch.
  Other Names: tongue plate
  Arms: Group A
Device: Fixed Face Mask — An extra-oral appliance used for treatment of maxillary deficiency in growing patients. It takes anchorage from the chin and forehead, has a fixed intra-oral appliance with an expansion screw and hooks for elastics that exert a force of 300 gr. It should be used 14 hours a day.
  Other Names: face mask
  Arms: Group B

SUMMARY:
A new fixed appliance will be used to transfer the tongue force during its physiological activity to advance the nasomaxillary complex; this method will be compared with the traditional method which uses a facemask with a fixed appliance in the mouth.

DETAILED DESCRIPTION:
The above method will be compared with traditional one which uses the facemask in combination with an intra-oral fixed appliance.

ELIGIBILITY:
Inclusion Criteria:

* Growing patients
* Class III with maxillary deficiency

Exclusion Criteria:

* Previous orthodontic treatment
* Uncooperative patients

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-04 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Cephalometric angles and clinical features | At least 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rahman Showkatbakhsh, Professor, Study Chair — Shaheed Beheshti dental school; Mohammad Behnaz, Principal Investigator — Shahid Beheshti Dental school
Locations (1):
- Shahid Beheshti Medical University, Tehran, Iran